CLINICAL TRIAL: NCT00241137
Title: A Study to Compare Treating Hypertension With Valsartan 160 MG to Valsartan 320 Mg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489H2301
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2006-06

CONDITIONS: Hypertension
Keywords: hypertension; valsartan
MeSH Terms: conditions — Hypertension | interventions — Valsartan

INTERVENTIONS:
Drug: valsartan

SUMMARY:
The purpose of this was to evaluate valsartan 320mg compared to valsartan 160 mg in terms of blood pressure reduction in a patient population of mild to moderate hypertensives

ELIGIBILITY:
Inclusion Criteria:

* • Male or female age between 18-80 years of age, inclusive

  * Diagnosed at enrollment (visits 2) to be mild to moderate hypertensive with a MSDBP >= 95 and =< 109 mmHg for non treated patients.
  * Previously treated patients should have a MSDBP =< 109 mmHg at visit 1 and a MSDBP >= 95 and =< 109 mmHg at visit 2.
  * Written informed consent to participate in the study prior to any study procedures
  * Ability to communicate and comply with all study requirements

Exclusion Criteria:

* Severe hypertension (grade 3 of WHO classification; >= 110 mmHg diastolic and/or >= 180 mmHg systolic).
* Malignant hypertension
* Inability to discontinue all prior anti-hypertensive medications safely for a period of 2 weeks, as required by the protocol.
* Known history of proteinuria (greater than 0.3 gram per day)
* Female patients who are not either post-menopausal for one year or surgically sterile, and who are not using effective contraceptive methods such as barrier method with spermicidal or an intra-uterine device. Oral contraceptive use is not allowed.
* Known Keith-Wagener grade III or IV hypertensive retinopathy.
* History of hypertensive encephalopathy or cerebrovascular accident at anytime prior to Visit 1.
* Transient ischemic cerebral attack during the last 12 months prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3790 (Actual)
Dates: Start 2003-09; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline diastolic blood pressure after 4 weeks

SECONDARY OUTCOMES:
Change from baseline systolic blood pressure after 4 weeks
Change from baseline diastolic and systolic blood pressure in patients with a diastolic blood pressure greater than or equal to 90 mmHg at randomization after 4 weeks
Adverse events and serious adverse events at each study visit for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceutical, Study Director — Novartis Pharmaceuticals
Locations (1):
- Investigative Centers, Germany